CLINICAL TRIAL: NCT05160129
Title: Connectomic Deep Brain Stimulation for Obsessive Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martijn Figee, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-00125; 1R01MH123542-01 (NIH)
Record Dates: First submitted 2021-11-17; First posted 2021-12-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: Deep Brain Stimulation (DBS); Obsessive Compulsive Disorder (OCD); Anterior Limb of Internal Capsule (ALIC); Circuit Modulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Circuit-selective DBS (Experimental): People suffering from severe obsessive-compulsive disorder (OCD)
  Interventions: Device: Selective focal stimulation of ALIC-pathways

INTERVENTIONS:
Device: Selective focal stimulation of ALIC-pathways — DBS will be applied selectively to different electrode contacts/ segments to evaluate clinical, behavioral, and electrocortical responses of specific pathways within the ALIC.

SUMMARY:
Deep brain stimulation (DBS) is an effective treatment for people suffering from severe obsessive-compulsive disorder (OCD) whose symptoms have failed to improve after years and multiple methods of intervention. An effective DBS target for OCD is the anterior limb of the internal capsule (ALIC) brain region. On average 60% of all OCD patients have a clinically significant response to ALIC DBS. However, ALIC DBS may become even more effective with the ability to predict which specific ALIC connections in the brain need to be stimulated for each individual OCD patient. This study therefore investigates personalized stimulation to the ALIC that allows for precise modulation of brain circuits associated with individual OCD symptoms. The study aims to specify the ideal anatomical target for ALIC DBS for maximum therapeutic benefit in each patient.

DETAILED DESCRIPTION:
To improve DBS for severe OCD, the anatomical specificity with which stimulation is delivered must be enhanced. In this study, patients will receive personalized and circuit specific stimulation to five target ALIC pathways based on pre-surgery brain scan analysis where patient-specific blueprints are created and used to determine implant location. Stimulation to the ALIC is delivered by directional segmented electrodes which are designed to deliver precise activation of circuits of interest and minimize excess tissue activation that can cause side effects. In this study, ALIC DBS will target white matter pathways, each having different cortical projections that affect different behavioral outputs, instead of traditional targeting. Each of these chosen pathways have been shown to be involved in the effects of ALIC DBS for OCD, but the results vary between studies.

The current study involves routine implantation of bilateral DBS leads into the ALIC brain region, which are connected to an internal pulse generator (IPG) device that is implanted under the skin near the collar bone and controls stimulation delivery. Before surgery, patients will receive a high definition 7T MRI brain scan to carefully plan the personalized lead implantation. Following surgery, patients will receive routine clinical visits for optimizing the DBS parameters and monitoring of clinical effects. As part of this study, patients will participate in EEG recordings at stimulation initiation and after 6 and 12 months. In addition, patients will complete behavioral paradigm testing bimonthly during stimulation of circuit-specific DBS contacts.

The goal of this study is to create a blueprint map of the brain that characterizes pathways that are found in effective treatment of OCD. This will be done by determining which pathways are activated by stimulation in different locations in ALIC and linking these locations with changes in task performance. This will allow for specification of the ideal anatomical target for DBS for OCD for maximum therapeutic benefit.

ELIGIBILITY:
All participants will receive ALIC DBS for OCD. DBS received a Humanitarian Device Exemption (HDE) in 2009 with an indication for bilateral stimulation of the ALIC as an adjunctive treatment to medications and as an alternative to anterior capsulotomy for treatment of chronic, severe, treatment-refractory OCD in adult patients who have failed at least three SSRIs. Additionally, more stringent criteria have been selected for defining treatment-resistance in this protocol, as indicated below.

INCLUSION CRITERIA:

* 18 years of age or older
* Primary psychiatric diagnosis of Obsessive-Compulsive Disorder (OCD, per DSM-5 criteria)
* Meets FDA Humanitarian Device Exemption (HDE) criteria for indication
* Has elected to receive clinically indicated DBS for OCD with a directional system outside of this research study, as determined by treating clinician(s) and per current clinical practice
* Minimum of a five-year history of treatment-refractory OCD with substantial functional impairment
* Failure of an adequate trial of at least three of the following SSRIs: Fluoxetine, Fluvoxamine, Citalopram, Escitalopram, Sertraline, Paroxetine
* Failure of an adequate trial of clomipramine
* Failure of an adequate trial of one or more of the aforementioned antidepressants in combination with at least one of the following augmentation agents: Haloperidol, Risperidone, Olanzapine, Quetiapine, Ziprasidone, Aripiprazole
* Failure of an adequate trial of Cognitive Behavioral Therapy (CBT), defined as 25 hours of documented exposure and response prevention (ERP) by an expert therapist
* Minimum score of 25 on the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) at preoperative baseline
* Ability to undergo preoperative MRI
* English proficiency
* Capacity to provide written informed consent
* Willing and able to comply with all device operation and study-related procedures

EXCLUSION CRITERIA:

* Ineligible or unwilling to receive ALIC DBS for OCD
* Contraindications for general anesthesia, neurosurgery, or an MRI scan
* Neurological disorder or other significant brain pathology, such as moderate / marked cerebral atrophy, stroke, tumor, epilepsy, or previous neurosurgical procedures (excluding cingulotomy, which may be permitted if not contraindicated in the opinion of implanting neurosurgeon)
* Unstable medical illness, chronic immunosuppression, and/or considerably reduced life-expectancy
* Conditions requiring anticoagulant therapy which cannot be discontinued for the perioperative period, as required
* Conditions requiring certain regular MRI scans or diathermy
* Currently implanted with a cardiac pacemaker / defibrillator or other implanted electrical device which may interfere with DBS stimulator or the function of which may be impacted by its implantation, in the opinion of evaluating neurosurgeon
* Other primary Axis I disorder or history of psychosis, such as schizophrenia, psychosis in the context of depressive or manic episode.
* Current or past history within the 6 months prior to DBS implantation of substance abuse or dependence (excluding nicotine and caffeine)
* Active suicidal ideation with intent, suicide attempt within the last six months, more than three suicide attempts within the last two years, or serious suicide risk as determined by the study psychiatrists
* Axis II disorders which, in the opinion of the study psychiatrist, may increases the risk of DBS to participants or cause study non-compliance
* Patients who lack the capacity to for proper device usage and maintenance, in the opinion of the research team
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Yale Brown Obsessive Compulsive Scale (Y-BOCS) | Pre-surgical baseline, monthly up to 12 months postoperative
  This scale measures change in OCD symptom severity. Full scale from from 0 - 40 with higher score indicating more severe symptoms.

SECONDARY OUTCOMES:
Investment Task | Pre-surgical baseline, bimonthly up to 12 months postoperative
  This computational investment task provides a measure of reward valuation by measuring decision making related to different reward conditions.
  Computational computer tasks: These behavioral tasks provide a measure of reward valuation, cognitive flexibility under conditions of uncertainty, and a measure of inhibitory control.
Reversal Task | Pre-surgical baseline, bimonthly up to 12 months postoperative
  This computational reversal task provides a measure of cognitive flexibility under conditions of uncertainty.
  Computational computer tasks: These behavioral tasks provide a measure of reward valuation, cognitive flexibility under conditions of uncertainty, and a measure of inhibitory control.
Stop Signal Task | Pre-surgical baseline, bimonthly up to 12 months postoperative
  This computational stop signal task provides a measure of inhibitory control by assessing stop-signal reaction time.
  Computational computer tasks: These behavioral tasks provide a measure of reward valuation, cognitive flexibility under conditions of uncertainty, and a measure of inhibitory control.
Tractography pathway activation models (Diffusion-weighted-imaging) | Baseline: Pre-surgery
  Data collected from MRI scans will be used to measure structural connectivity in the brain (i.e., white matter pathways) that is used for surgical planning.
Deep brain stimulation evoked potentials (EEG) | postoperative months 0, 6, 12
  Evoked potentials provide a measure of electrophysiological, effective connectivity in the brain. Alpha, beta, theta, gamma and delta bandwidths will be assessed.
Change in Beck Depression Inventory (BDI) | Pre-surgical baseline, monthly up to 12 months postoperative
  This scale indicates the presence and severity of depressive symptoms. Full scale from 0 to 63 , with higher score indicating more severe depression.
Change in Beck Anxiety Inventory (BAI) | Pre-surgical baseline, monthly up to 12 months postoperative
  This scale measures severity of anxiety symptoms. Full scale from 0 to 63, with higher score indicating more severe anxiety.
Change in Barratt Impulsiveness Scale (BIS-11) | Pre-surgical baseline, monthly up to 12 months postoperative
  This is a clinical measure of impulsivity. Full scale from 30 -120, with a higher score indicating greater impulsivity.
Change in Young Mania Rating Scale (YMRS) | Pre-surgical baseline, monthly up to 12 months postoperative
  This scale measures the presence and severity of mania. Full scale from 0 - 60, with higher scores indicating more severe mania.
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) | Pre-surgical baseline, monthly up to 12 months postoperative
  This scale measures risk of suicide on multiple dimensions, scored by answering "yes or no" questions where answers of "yes" may indicate risk. Full range from 0 to 9, with higher score indicating higher intensity suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Figee, Principal Investigator — Icahn School of Medicine and Mount Sinai; Ki Sueng Choi, Principal Investigator — Icahn School of Medicine and Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. To achieve aims in the approved proposal. Proposals should be directed to Sonia.olson@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website.